CLINICAL TRIAL: NCT04347070
Title: Implementation of Physiotherapy on COVID-19 Patients in Intensive Care Units : a Retrospective, Multicentric, International Study
Brief Title: Implementation of Physiotherapy on COVID-19 Patients in ICU
Acronym: PHYSIO-COVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Société espagnole de pneumologie (SEPAR) (Unknown); Societe française de kinésithérapie en réanimation (SKR) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0175
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Sars-CoV2; COVID-19
Keywords: COVID-19; Physiotherapy; implementation; critical care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients accepted in ICU diagnosed with COVID-19: Patients accepted in ICU diagnosed with COVID-19
  Interventions: Other: Phsyiotherapy

INTERVENTIONS:
Other: Phsyiotherapy — To observe if patients with COVID-19 benefice of physiothersapy, which kind and how many time

SUMMARY:
Despite new charachersitics of COVID-19 patients, critical care implementation seems to be similar to those with Acute Respiratory Distress Syndrome (ARDS) in intensive care units (ICU).

Regarding the initial gravity of these patients, sedation and neuromuscular blockers are usually administrated, increasing the risk to develope an ICU-acquired weakness which is directly correlated to morbi-mortality and a burden during recovery.

Respiratory symptoms are mostly related to dyspnoea and non-productive cough, with only 33% of COVID-19 patient having a bronchial hypersecretion ; consequently, chest physiotherapy is only implemented in after case-by-case evaluation.

This unprecedented situation requires to identify how physiotherapy is being implemented in COVID-19 patients in ICU.

This retrospective, multicentric study aims to identify the charactheristics of physiotherapy (type and time spent) implemented in Argentina, Belgium, Chili, France, Italy and Spain

DETAILED DESCRIPTION:
* Demographics data : hospitalisation date, ICU date, COVID+ date, extubation date, discharge date, mortality
* ICU data : ventilatory mode, type of physiotherapy implemented (early rehabilitation, chest physiotherapy, time spent (minutes), number of interventions per day.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Patient admitted in ICU
* Patient with COVID-19 diagnosis

Exclusion criteria:

- Explicite denie to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU with COVID-19 will be eligible
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Time of physiotherapy | 1 day
  Time of physiotherapy (minutes)
Time of physiotherapy | 3 day
  Time of physiotherapy (minutes)
Time of physiotherapy | 7 day
  Time of physiotherapy (minutes)

SECONDARY OUTCOMES:
Type of physiotherapy implemented | 1 day
  Type of physiotherapy , early rehabilitation or chest phsyitoherapy
Type of physiotherapy implemented | 3 day
  Type of physiotherapy , early rehabilitation or chest phsyitoherapy
Type of physiotherapy implemented | 7 day
  Type of physiotherapy , early rehabilitation or chest phsyitoherapy

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Martinez-Alejos, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC